CLINICAL TRIAL: NCT00414531
Title: Investigations on Differences in Atorvastatin Metabolites Ratios as a Diagnostic Tool in Detecting Atorvastatin Induced Myotoxicity
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Oslo School of Pharmacy (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: Single | Purpose: Diagnostic
Other Study IDs: AVALIP05
Record Dates: First submitted 2006-12-20; First posted 2006-12-21 (Estimated); Last update posted 2014-12-03 (Estimated); Status verified 2009-08

CONDITIONS: Myotoxicity of Atorvastatin Treatment
MeSH Terms: interventions — Atorvastatin

STUDY DESIGN:
Who Masked: Investigator

ARMS (1):
- SIM (Other): Patients diagnosed to have or not to have Statin induced Myopathy
  Interventions: Drug: Atorvastatin

INTERVENTIONS:
Drug: Atorvastatin — 20 to 80 mg per day

SUMMARY:
The primary objective of the study is to investigate the ratios of p-hydroxyatorvastatin to atorvastatin in patients receiving atorvastatin treatment, who experience muscle adverse events, to elucidate whether differences in this ratio might have a positive or negative predictive value in diagnosing atorvastatin muscle toxicity.

DETAILED DESCRIPTION:
The primary objective of the study is to investigate the ratios of p-hydroxyatorvastatin to atorvastatin in patients receiving atorvastatin treatment, who experience muscle adverse events, to elucidate whether differences in this ratio might have a positive or negative predictive value in diagnosing atorvastatin muscle toxicity. If this is shown, measurements of atorvastatin metabolites from patients experiencing muscle adverse events might be a valuable diagnostic tool to diagnose myopathy associated with statin treatment. The primary endpoint cut off level for present myotoxicity has been set to a ratio of p-hydroxyatorvastatin /atorvastatin of 0.15 from the previously performed pilot study (Unpublished data, Herman M et al). Values at or above this ratio will be considered as clinical significant indicia of statin related myopathy.

Secondary objectives include descriptively investigation of drug to metabolite cut off ratio for atorvastatin lactone/atorvastatin. Whether other cut off values, both for p-hydroxyatorvastatin as well as for atorvastatin lactone, give more precise identification of patients that are experiencing statin related myopathy compared to controls will also be investigated.

Explorative objectives of the study are to investigate possible in vitro phenotypic differences in isolated muscle cells from patients experiencing muscle toxicity compared to patients not experiencing muscle toxicity. If there are genetic differences between patients experiencing myotoxicity and those not, this difference is likely to show as phenotypic differences in in vitro studies of isolated muscle cells. If such phenotypic differences are present in vitro possible mechanistic causes will be further investigated.

ELIGIBILITY:
Inclusion Criteria:

* Suspected atorvastatin induced muscle adverse events.
* Signed informed consent.
* 18 years of age or older.
* Able to donate blood samples.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Actual)
Dates: Start 2005-05; Primary Completion 2009-06 (Actual); Study Completion 2009-06 (Actual)

PRIMARY OUTCOMES:
ratio of p-hydroxyatorvastatin to atorvastatin vs. myopathy | march 2009

SECONDARY OUTCOMES:
ratio of atorvastatin lactone to atorvastatin vs. myopathy | march 2009

CONTACTS AND LOCATIONS:
Overall Officials: Anders Åsberg, Ph.D., Study Director — Universtiy of Oslo
Locations (1):
- Rikshospitalet-Radiumhospitalet HF, Lipid clinic, Oslo, Norway

REFERENCES:
- [Derived] Skottheim IB, Bogsrud MP, Hermann M, Retterstol K, Asberg A. Atorvastatin metabolite measurements as a diagnostic tool for statin-induced myopathy. Mol Diagn Ther. 2011 Aug 1;15(4):221-7. doi: 10.1007/BF03256413. PMID 21815705